CLINICAL TRIAL: NCT02795156
Title: Phase II Study to Evaluate the Activity of Commercially Available Molecularly Matched Targeted Therapies in Selected Tumor Types Based on Genomic Alterations
Brief Title: Study Assessing Activity of Molecularly Matched Targeted Therapies in Select Tumor Types Based on Genomic Alterations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Foundation Medicine (Industry); Boehringer Ingelheim (Industry); Bayer (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI PRO 10
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Carcinoma; Urothelial Carcinoma; Gastrointestinal Carcinoma, Non-colon; Upper Aerodigestive Tract Carcinoma
Keywords: regorafenib; afatinib; targeted therapy; cabozantinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell | interventions — Afatinib; regorafenib; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): Patients with non-small cell lung cancer who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Interventions: Drug: Afatinib; Drug: Regorafenib; Drug: Cabozantinib
- Arm 2 (Experimental): Patients with urothelial carcinoma who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Interventions: Drug: Afatinib; Drug: Regorafenib; Drug: Cabozantinib
- Arm 3 (Experimental): Patients with non-colon gastrointestinal cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Interventions: Drug: Afatinib; Drug: Regorafenib; Drug: Cabozantinib
- Arm 4 (Experimental): Patients with upper aerodigestive tract cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Interventions: Drug: Afatinib; Drug: Regorafenib; Drug: Cabozantinib

INTERVENTIONS:
Drug: Afatinib — 40 mg orally once daily for each 28-day cycle. Treatment will continue until disease progression or intolerable toxicity or other reason for discontinuation up to 45 months.
  Other Names: Gilotrif
Drug: Regorafenib — 160 mg orally once daily for the first 21 days of each 28-day cycle. Treatment will continue until disease progression or intolerable toxicity or other reason for discontinuation up to 45 months.
  Other Names: Stivarga
Drug: Cabozantinib — 60 mg orally once daily for each 28-day cycle. Treatment will continue until disease progression or intolerable toxicity or other reason for discontinuation up to 45 months.
  Other Names: Cabometyx

SUMMARY:
With the increased availability of next-generation sequencing, oncologists are starting to incorporate genomic profiling into routine care of cancer patients. If a genomic alteration is identified during profiling, it could help guide the choice of therapy and improve treatment outcomes. This study will examine the anti-tumor activity of selected commercially available molecularly matched targeted therapies in patients who have failed first-line treatment for one of the following tumor types: non-small cell lung cancers; urothelial cancer; non-colon gastrointestinal cancers, and upper aerodigestive tract cancer.

DETAILED DESCRIPTION:
This four-arm pilot phase II study will evaluate the preliminary antitumor activity of selected commercially available molecularly matched targeted therapies in patients who have failed first line treatment for one of the following tumor types:

1. non-small cell lung cancer,
2. urothelial carcinoma,
3. non-colon gastrointestinal cancers, and
4. upper aerodigestive tract cancers (lip, tongue, salivary glands, gum, mouth, oral cavity, tonsils, oropharynx, nasopharynx, nasal cavity, sinus, and larynx tumors).

Approximately 160 patients (40 per tumour type) are planned for enrollment. Consideration for enrollment will be based on results from profiling with next-generation sequencing technology that was performed outside of the protocol. Eligible patients will receive one of the FDA-approved targeted agents at the recommended dose. The treating physician will decide which targeted agent to prescribe based on the genomic alterations per tumor type and the targets listed in the package insert for each agent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically or cytologically confirmed diagnosis of one of the following tumor types whose disease has progressed following one line of standard therapy and/or for which no standard treatment is available that has been shown to prolong survival:

   1. Non-small cell lung cancer
   2. Urothelial carcinoma
   3. Non-colon gastrointestinal cancers (including hepatobiliary, pancreatic, and gastroesophageal tumors)
   4. Upper aerodigestive tract cancers (including lip, tongue, salivary gland, gum, oral cavity, mouth, tonsils, oropharynx, nasopharynx, nasal cavity, sinus, and larynx tumors)
2. Patients must have a predefined genomic alteration that can be targeted with any of the FDA-approved targeted agents used in this study.
3. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Age greater than or equal to 18 years.
6. Adequate hematologic function defined as:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Platelets ≥75,000/μL
7. Adequate liver function defined as:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x the upper limit of normal (ULN) or ≤ 5.0 X ULN if liver metastases present
   * Total bilirubin ≤1.5 x ULN (unless the patient has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin)
8. Adequate renal function defined as serum creatinine ≤1.5 x the upper limit of normal OR measured or calculated creatinine clearance ≥50 mL/min for patients with creatinine levels greater than or equal to 1.5 x the upper limit of normal.
9. Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to receive either regorafenib or afatinib provided that their medication dose and INR/PTT are stable. Close monitoring is mandatory if the patient is receiving anticoagulants. If values are above the therapeutic range the anticoagulant doses should be modified and assessments should be repeated until stable.
10. Male patients with female partners of childbearing potential and women patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 90 days following last dose of study drug(s). Male patients must also refrain from donating sperm during their participation in the study and for 90 days after the last dose of study drug.
11. Willingness and ability to comply with study and follow-up procedures.
12. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Two or more prior chemotherapy regimens in the metastatic setting.
2. Most recent chemotherapy ≤ 3 weeks and > Grade 1 chemotherapy-related side effects, with the exception of neuropathy (> grade 2 excluded) and alopecia.
3. Use of a study drug or targeted therapy ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of study treatment. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of study treatment is required.
4. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
5. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
6. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks prior to study entry and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy. Enzyme-inducing anticonvulsants are contraindicated.
7. Pregnant or lactating
8. Acute or chronic liver, renal, or pancreas disease.
9. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy.
10. Any of the following cardiac diseases currently or within the last 6 months:

    * Unstable angina pectoris
    * Congestive heart failure (New York Heart Association (NYHA) ≥ Grade 2
    * Acute myocardial infarction
    * Conduction abnormality not controlled with pacemaker or medication
    * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
    * Valvular disease with significant compromise in cardiac function
11. Inadequately controlled hypertension.
12. Thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of treatment.
13. Evidence or history of bleeding diathesis or coagulopathy; any haemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of treatment.
14. For patients receiving cabozantinib only: Do not administer cabozantinib to patients that have high risk or at high risk for severe haemorrhage. Examples include:

    1. The patient has radiographic evidence of cavitating pulmonary lesion(s).
    2. The patient has tumor invading or encasing any major blood vessels.
    3. The patient has had hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment.
    4. The patient has experienced clinically significant GI bleeding within 6 months of the first dose of study treatment.
    5. The patient has experienced any other signs indicative of pulmonary hemorrhage within 3 months of the first dose of study treatment.
15. For patients receiving cabozantinib only: Do not administer cabozantinib to patients that have high risk or at high risk of perforation or fistula:

    1. The patient has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    2. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.
    3. The patient has pre-existing fistula of head and neck area. Note: Treatment areas should be healed with no sequelae from prior radiation therapy that would predispose to fistula formation.
    4. The patient has pre-existing osteonecrosis of the jaw.
16. Concomitant anticoagulation at therapeutic doses with oral anticoagulants or platelet inhibitors. [Patients receiving cabozantinib only]
17. Note: Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (< 1 mg/day), and low dose, low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 12 weeks before randomization, and who have had no complications from a thromboembolic event or the anticoagulation regimen.Presence of a non-healing wound, non-healing ulcer, or bone fracture.
18. Patients with phaeochromocytoma.
19. Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
20. Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C.
21. Presence of other active cancers unless indolent and not requiring therapy. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma are eligible, as are patients with history of non-melanoma skin cancer.
22. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, III, MD, Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Research Medical Center - HCA Midwest, Kansas City, Missouri
  - Tennesse Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients with non-small cell lung cancer who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally once daily for each 28-day cycle
  regorafenib: 160 mg orally once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg orally once daily for each 28-day cycle
- Arm 2: Patients with urothelial carcinoma who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Afatinib: 40 mg orally once daily for each 28-day cycle
  Regorafenib: 160 mg orally once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg orally once daily for each 28-day cycle
- Arm 3: Patients with non-colon gastrointestinal cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  Afatinib: 40 mg orally once daily for each 28-day cycle
  Regorafenib: 160 mg orally once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg orally once daily for each 28-day cycle
- Arm 4: Patients with upper aerodigestive tract cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally once daily for each 28-day cycle
  regorafenib: 160 mg orally once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg orally once daily for each 28-day cycle
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 39 | 10 | 42 | 9
Completed | 0 | 0 | 0 | 0
Not Completed | 39 | 10 | 42 | 9
Not completed — Progressive Disease | 22 | 7 | 34 | 7
Not completed — Adverse Event | 13 | 2 | 3 | 2
Not completed — Death | 1 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Patients with non-small cell lung cancer who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally (p.o.) once daily for each 28-day cycle
  regorafenib: 160 mg p.o. once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg p.o. once daily for each 28-day cycle
- Arm 2: Patients with urothelial carcinoma who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally (p.o.) once daily for each 28-day cycle
  regorafenib: 160 mg p.o. once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg p.o. once daily for each 28-day cycle
- Arm 3: Patients with non-colon gastrointestinal cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally (p.o.) once daily for each 28-day cycle
  regorafenib: 160 mg p.o. once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg p.o. once daily for each 28-day cycle
- Arm 4: Patients with upper aerodigestive tract cancers who have failed first line treatment may receive either regorafenib (Stivarga), afatinib (Gilotrif), or cabozantinib (Cabometyx) at the recommended dose level, depending on their specific genomic alterations.
  afatinib: 40 mg orally (p.o.) once daily for each 28-day cycle
  regorafenib: 160 mg p.o. once daily for the first 21-days of each 28-day
  Cabozantinib: 60 mg p.o. once daily for each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 39 | 10 | 42 | 9 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 12 | 5 | 28
  >=65 years | 30 | 8 | 30 | 4 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 3 | 13 | 1 | 42
  Male | 14 | 7 | 29 | 8 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 0 | 5
  White | 35 | 10 | 39 | 9 | 93
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 10 | 42 | 9 | 100

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Each Arm Receiving Targeted Therapy Based on Relevant Genomic Alterations
Description: ORR is defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR), i.e., two CRs and/or PRs at least 4 weeks apart, according to the RECIST v1.1 criteria. CR=disappearance of all target and non-target lesions. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: every 8 weeks until tumor progression or treatment discontinuation, up to 45 months.
Population: All enrolled patients are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 39 | 10 | 42 | 9
percentage of participants | 10.3 [2.87 to 24.22] | 0 [NA to NA] — No participants in this arm met the definition of Overall Response Rate. Confidence interval can't be calculated. | 7.1 [1.5 to 19.48] | 0 [NA to NA] — No participants in this arm met the definition of Overall Response Rate. Confidence interval can't be calculated.

2. Secondary Outcome: Clinical Benefit Rate in Each Arm Receiving Targeted Therapy Based on Relevant Genomic Alterations
Description: Clinical Benefit Rate (CBR) is defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR) or stable disease (SD) ≥ 6 months according to RECIST v1.1. Confirmed response is defined as two CRs and/or PRs at least 4 weeks apart, according to the RECIST v1.1 criteria. CR=disappearance of all target lesions. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease= Neither sufficient shrinkage to qualify for PR nor sufficient increase of 20% in the sum of diameters or presence of a new lesion to qualify for progressive disease (PD), taking as reference the smallest (nadir) sum of diameters since the treatment started.
Time Frame: Every 8 weeks until tumor progression or treatment discontinuation, up to 45 months
Population: All enrolled participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 39 | 10 | 42 | 9
percentage of participants | 15.4 [5.86 to 30.5] | 0 [NA to NA] — No participants met the definition of Clinical Benefit Rate. There is no confidence interval to be calculated. | 21.4 [10.3 to 36.8] | 11.1 [.28 to 48.2]

3. Secondary Outcome: Time to Treatment Failure (TTF) in Each Arm Receiving Targeted Therapy Based on Relevant Genomic Alterations
Description: Time to treatment failure is measured from the first day of treatment until the patient is removed from study for toxicity, disease progression per RECIST v1.1, patient choice, or death. Progressive disease (PD) per RECIST v1.1 is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum since the treatment started, or the appearance of one or more new lesions. Requires not only 20% increase, but absolute increase of a minimum of 5 mm over the sum.
Time Frame: Every 8 weeks until tumor progression or treatment discontinuation, up to 45 months
Population: All enrolled participants were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 39 | 10 | 42 | 9
months | 2.1 [1.6 to 2.8] | 1.8 [1.1 to 1.9] | 1.9 [1.8 to 3.5] | 2.0 [1.0 to 4.3]

4. Secondary Outcome: Progression-Free Survival in Each Arm Receiving Targeted Therapy Based on Relevant Genomic Alterations
Description: Progression Free Survival (PFS) is defined as the time from the first day of study drug administration (Day 1) to disease progression as defined by the RECIST v1.1, or death on study. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment. Progressive disease (PD) per RECIST v1.1 is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum since the treatment started, or the appearance of one or more new lesions. Requires not only 20% increase, but absolute increase of a minimum of 5 mm over the sum.
Time Frame: Every 8 weeks until tumor progression or treatment discontinuation, up to 45 months
Population: All enrolled participants were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 39 | 10 | 42 | 9
months | 3.2 [2.7 to 4.4] | 1.9 [1.5 to 3.3] | 3.1 [2.3 to 4.2] | 2.8 [1.8 to 8.6]

ADVERSE EVENTS:
Time Frame: Serious and/or other adverse events were assessed from the date of first dose to 30 days after last dose of study treatment, up to 45 months. All-Cause Mortality was monitored from date of consent up until progression of disease or death, up to 45 months.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 14/39 | 1/10 | 13/42 | 3/9
Serious Adverse Events (participants affected / at risk) | 16/39 | 6/10 | 14/42 | 5/9
Other Adverse Events (participants affected / at risk) | 39/39 | 10/10 | 41/42 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=39) | Arm 2 (N=10) | Arm 3 (N=42) | Arm 4 (N=9)
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=39) | Arm 2 (N=10) | Arm 3 (N=42) | Arm 4 (N=9)
Diarrhoea (Gastrointestinal disorders) | 17 | 10 | 22 | 3
Nausea (Gastrointestinal disorders) | 20 | 7 | 18 | 1
Vomiting (Gastrointestinal disorders) | 11 | 5 | 10 | 0
Constipation (Gastrointestinal disorders) | 9 | 2 | 8 | 3
Stomatitis (Gastrointestinal disorders) | 9 | 2 | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 6 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 17 | 2 | 17 | 3
Dehydration (Metabolism and nutrition disorders) | 16 | 8 | 12 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 19 | 7 | 20 | 4
Mucosal inflammation (General disorders) | 5 | 4 | 5 | 1
Asthenia (General disorders) | 3 | 0 | 3 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1 | 2
Chills (General disorders) | 1 | 2 | 2 | 0
Pain (General disorders) | 2 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 5 | 0
Gait disturbance (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 12 | 2 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 6 | 1
Blood bilirubin increased (Investigations) | 4 | 0 | 7 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 5 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 7 | 0
Platelet count decreased (Investigations) | 3 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2 | 0
Blood albumin decreased (Investigations) | 2 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Protein total increased (Investigations) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 1 | 5 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 0 | 5 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 4 | 0
Tremor (Nervous system disorders) | 1 | 1 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 3 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 1
Rash pustular (Infections and infestations) | 2 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 7 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 3 | 0
Depression (Psychiatric disorders) | 4 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 2 | 5 | 0
Hypertension (Vascular disorders) | 2 | 1 | 4 | 0
Hot flush (Vascular disorders) | 0 | 1 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 4 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 2 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0
Blindness (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Stent placement (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02795156/Prot_SAP_000.pdf